CLINICAL TRIAL: NCT03618940
Title: Developing, Implementing and Evaluating Intervention Module on Preventing Fire, Burns and Scalds Injury Among Children Ages 7 to 11 Years In Sentul, Kuala Lumpur
Brief Title: Module on Preventing Fire, Burns and Scalds Injury Among Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Putra Malaysia (Other)
Collaborators: Honeywell Home Solutions USA (Unknown); Safe Kids Worldwide USA (Unknown)
Responsible Party: Principal Investigator, Assoc Prof Dr Kulanthayan K.C. Mani, principal investigator, Universiti Putra Malaysia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Child Fire and Burn Injury
Record Dates: First submitted 2018-07-16; First posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Burn Injury
Keywords: fire; burn injury; children; scalds
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- School-based educational intervention (Experimental): 1. assessed for knowledge and attitude on burn injury prevention
  2. underwent the School-based educational intervention
  3. impact evaluation
  4. Output evaluation 3 months after School-based educational intervention
  Interventions: Behavioral: Knowledge and Attitude on burn prevention

INTERVENTIONS:
Behavioral: Knowledge and Attitude on burn prevention — 1.Introduction to Home Safety
  2 Fire Safety & Burn Safety (Cooking Safety, Safety around Motorcycle Exhaust &First Aid for Minor Burns
  3 Electrical Safety (Safety around Electrical & Appliances & Outlets)
  4 Firecrackers Safety (Safety around Firecrackers & Open Flames)
  5. Escaping from Fire (Escaping from Fire, Calling for Help, Stop, Drop & Roll, Emergency Calling Number (By Fire Department Kuala Lumpur), Show equipment/gear that firefighters use, Demonstrate how to use the fire extinguisher, Crawl low in smoke

SUMMARY:
The main aim of this intervention study is to test the hypothesis if school based educational intervention program will significantly improve the knowledge of primary school student on childhood burn prevention in Kuala Lumpur. The secondary aim the evaluate the association of demographics background, burn injury history with knowledge on burn. The study was conducted in 12 primary school in Kuala Lumpur from 1st January 2015 to 31st December 2017 in three different phases.

DETAILED DESCRIPTION:
According to World Health Organization data, approximately 10% of all unintentional injury deaths are due to fire-related burns. In Malaysia, burn represent about 5.6% (745 cases) of all injuries among children. As childhood burn was not considered as a child health problem comparing to other childhood illnesses, parents and children tends to have less priority in overcome this issue. This highlights the need to transfer the knowledge especially to the children on the burn prevention. By implementing this module on preventing fire, burns and scalds injury among children, knowledge on main causes of burns and their immediate management can be improved at young age.

ELIGIBILITY:
Inclusion Criteria:

* Students who are aged 7 till 11 years old
* Parent or guardian of each selected student above

Exclusion Criteria:

● Students under special needs class (Pendidikan Khas)

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2335 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Improve the knowledge on burn prevention among children | through study completion, an average of 2 year
  Educational intervention was conducted to improve the knowledge on burn prevention among children. The intervention uses Module on Preventing Fire, Burns and Scalds which consist of 5 main topics;
  1. Introduction to Home Safety
  2. Fire Safety & Burn Safety
  3. Electrical Safety
  4. Firecrackers Safety
  5. Escaping from Fire
  The knowledge on burn prevention was assessed using questionnaire before and after intervention. The total score of knowledge was further categorized into poor moderate and good.
  The change in mean score of knowledge was assessed using paired-t test and ANCOVA test
Improve the attitude on burn prevention among children | through study completion, an average of 2 year
  Educational intervention was conducted to improve the attitude on burn prevention among children. The intervention uses Module on Preventing Fire, Burns and Scalds
  The attitude on burn prevention was assessed using questionnaire before and after intervention. The total score of attitute was further categorized into poor moderate and good.
  The change in mean score of attitude was assessed using paired-t test and ANCOVA test

SECONDARY OUTCOMES:
Socio-demographic characteristic was associated with knowledge on burn prevention among children | first year of the study (1 year)
  A structured questionnaire was used to assess the socio-demographic characteristics of the children (age, gender, ethnicity, family income, educational background of parents, type of residential and number of siblings)
  the association between socio-demographic characteristics and knowledge on burn prevention among children was tested using ANOVA and Regression analysis
Socio-demographic characteristic was associated with attitude on burn prevention among children | first year of the study (1 year)
  A structured questionnaire was used to assess the socio-demographic characteristics of the children (age, gender, ethnicity, family income, educational background of parents, type of residential and number of siblings)
  the association between socio-demographic characteristics and attitude on burn prevention among children was tested using ANOVA and Regression analysis
Burn injuries was associated with knowledge on burn prevention among children | first year of the study (1 year)
  A structured questionnaire was used to gather information of burn injuries (history of burn, duration, location, severity)
  the association between burn injury and knowledge on burn prevention among children was tested using ANOVA and Regression analysis
Burn injuries was associated with attitude on burn prevention among children | first year of the study (1 year)
  A structured questionnaire was used to gather information of burn injuries (history of burn, duration, location, severity)
  the association between burn injury and attitude on burn prevention among children was tested using ANOVA and Regression analysis
Educational Module on Preventing Fire, Burns and Scalds Injury will be developed based on five main issues identified in pre-intervention phase | second year of the study (24 months)
  Education module will developed based on 5 main topics as identified in phase I (pre-intervention);
  1. Introduction to Home Safety
  2. Fire Safety & Burn Safety
  3. Electrical Safety
  4. Firecrackers Safety
  5. Escaping from Fire
  The module will be used as teaching materials on on Preventing Fire, Burns and Scalds Injury in primary school

CONTACTS AND LOCATIONS:
Locations (1):
- Primary Schools in Sentul District, Sentul, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided
plan to share the data for international collaboration or policy making